CLINICAL TRIAL: NCT01590368
Title: A Comparative Wear Test of Two Adhesives on the Unilect ™ Biotab Short Term Monitoring Electrode
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: UM-1015-12-U365
Record Dates: First submitted 2012-05-01; First posted 2012-05-02 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Marketed electrode (Other): The currently marketed electrodes using the current CE marked adhesive
  Interventions: Device: Marketed electrode
- Modified hydrogel (Active Comparator): Electrodes with the new modified adhesive - the "test" electrodes
  Interventions: Device: Modified "test" electrode

INTERVENTIONS:
Device: Marketed electrode — 12 electrodes will be placed on the subject for an ECG reading to be taken
  Arms: Marketed electrode
Device: Modified "test" electrode — 12 electrodes with modified adhesive will be placed on the subject to allow an ECG reading to be taken
  Arms: Modified hydrogel

SUMMARY:
It is hypothesised that the adhesion of electrodes and acceptability of the Electrocardiogram (ECG) trace is comparable between the two groups (marketed and test products) after 30 minutes (the intended period of use) of the electrodes.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Be a healthy volunteer and be over 18 years of age
* Willing to attend two scheduled visits for application and removal of the device and adverse event review
* Have healthy unbroken skin

Exclusion Criteria:

* Subjects with a history of sensitivity to any one of the components of the device being studied
* Subjects who have a history of skin related disorders to the chest.
* Subjects who are actively involved in the development, manufacturing, quality and marketing of Unomedical electrodes
* Subjects who have any other medical condition which, according to the investigator justifies exclusion from the study
* Subjects who have any current cardiac conditions that may lead to an abnormal ECG trace

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Product Performance : Remain in place | 30 minutes
  Ability to remain in place for a duration of 30 minutes (as per intended use)
Product Performance: Perform | 30 minutes
  Ability of the electrodes to perform after a duration of 30 minutes of wear (ECG tracing) as per intended use.

SECONDARY OUTCOMES:
Safety: Adverse Events | 2 days
  Safety will be evaluated by the nature and frequency of adverse events, (including condition of the skin under the electrodes using the Skin Irritation Scale (Appendix 4)) and ease of removal
Skin Rating | 2 days
  Condition of the skin under the electrodes using the Skin Irritation Scale

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A Schofield, Principal Investigator — North Cheshire Hospital